CLINICAL TRIAL: NCT06344338
Title: Application of Targeting Transcranial Direct Current Stimulation (tDCS) Stimulation in the Treatment of Refractory Status Epilepticus
Brief Title: Application of tDCS Stimulation in Controlling Refractory Status Epilepticus
Acronym: tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Weibi Chen, associate professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z211100002921030
Record Dates: First submitted 2024-03-19; First posted 2024-04-03 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Refractory Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The patients who meet the eligibility requirements will be randomized in a 1:1 ratio to undergo targeting tDCS stimulation (up to 10 times) or sham stimulation
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS treatment group (Experimental): In the real tDCS stimulation group, direct cathodal current at 2 mA was delivered by a tDCS device over the seizure onset zone. Anode was on the contralateral forehead. Treatment was for 20 min, repeated twice in a day, then again over the next few days. The maximum number of stimuli required to terminate the status epilepticus should not exceed 10.
  Interventions: Device: tDCS stimulation
- TDCS sham-stimulation group (Sham Comparator): The duration and frequency of tDCS treatments in the sham-stimulation group are the same as those in the treatment group, but the tDCS device is not active during the 20 minutes of sham-stimulation.
  Interventions: Device: TDCS sham-stimulation

INTERVENTIONS:
Device: tDCS stimulation — In the real-stimulation group, Treatment was for 20 min, repeated twice in a day, then again over the next few days. The maximum number of stimuli required to terminate the status epilepticus should not exceed 10. In the sham-stimulation group, The duration and frequency of tDCS are the same as those in the treatment group, but the tDCS device is not active during the 20 minutes of sham-stimulation
  Arms: tDCS treatment group
Device: TDCS sham-stimulation — TDCS sham-stimulation
  Arms: TDCS sham-stimulation group

SUMMARY:
The purpose of the study is to assess the efficacy and safety of targeting tDCS stimulation for treatment of Refractory status epilepticus

DETAILED DESCRIPTION:
After being informed about the study and potential risks, the recruited patients, giving written informed consent, will be determined of the eligibility for study entry. The patients who meet the eligibility requirements will be randomized in a 1:1 ratio to undergo targeting tDCS stimulation (up to 10 times) or sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 80 year-old with Gender unlimited,
* Suitable for EEG monitoring;
* Clinical diagnosis of Refractory status epilepticus (status epilepticus that cannot be controlled by two types of antiepileptic drugs and at least one anesthetic);
* Informed consent to participate in this study was obtained from the participants or their surrogates

Exclusion Criteria:

* Unstable vital signs (systolic blood pressure<90mmHg, heart rate<60 beats/min, pulse oxygen saturation<90%);
* Having severe skull injury/defect or medical equipment implanted in the head;
* Pregnancy;
* With any implantable electronic instrument (including pacemakers, vagus nerve stimulators) or metal implanted devices.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with status epilepticus termination between tDCS treatment group and tDCS sham--stimulation group as assessed by Salzburg Consensus Criteria for Non-Convulsive Status Epilepticus | through study completion, an average of 1 year
  Outcomes will be assessed by clinical observation and EEG evaluation before 10 times of tDCS stimulation between both groups

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events between tDCS treatment group and tDCS sham--stimulation group | through study completion, an average of 1 year
  Treatment-emergent adverse events will be assessed by clinical observation between tDCS treatment group and tDCS sham--stimulation group

CONTACTS AND LOCATIONS:
Overall Officials: Weibi Chen, Dr, Study Director — Xuanwu Hospital, Beijing; Jiaqing Yan, Dr, Principal Investigator — College of Electrical and Control Engineering, North China University of Technology
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
This study is an exploratory study, and the important information is the signal analysis of electroencephalogram (EEG). However, these data were huge, which makes it difficult to export, save and upload. Meanwhile, the EEG data also require special softwares to read after being exported

REFERENCES:
- [Result] Fisher RS, McGinn RJ, Von Stein EL, Wu TQ, Qing KY, Fogarty A, Razavi B, Venkatasubramanian C. Transcranial direct current stimulation for focal status epilepticus or lateralized periodic discharges in four patients in a critical care setting. Epilepsia. 2023 Apr;64(4):875-887. doi: 10.1111/epi.17514. Epub 2023 Feb 7. PMID 36661376
- [Result] Rezakhani S, Amiri M, Weckhuysen S, Keliris GA. Therapeutic efficacy of seizure onset zone-targeting high-definition cathodal tDCS in patients with drug-resistant focal epilepsy. Clin Neurophysiol. 2022 Apr;136:219-227. doi: 10.1016/j.clinph.2022.01.130. Epub 2022 Feb 3. PMID 35217351